CLINICAL TRIAL: NCT06215703
Title: Optimizing Music-based Interventions for Stroke: a Mechanistic Crossover Study of the Effects of Music Improvisation and Live Accompaniment on Motor, Autonomic, and Neural Response During a Music Playing Task Among Survivors of Stroke and Matched Healthy Control Participants
Brief Title: Optimizing Music-Based Interventions for Stroke
Acronym: OptiMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-01380
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: stroke; healthy; music; MRI
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A 2x2 crossover design will be used such that each participant will complete all music playing conditions, including: (1) with or without improvisation and (2) with or without live accompaniment. Participants will be randomized to one of four condition orders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Order 1 (Experimental): Participants randomized to Order 1 will complete the four music playing tasks in the following order: (1) No improvisation (maintain beat), no live accompaniment (recorded accompaniment); (2) Improvisation, no live accompaniment (recorded accompaniment); (3) No Improvisation (maintain beat), live accompaniment; (4) Improvisation, live accompaniment.
  Interventions: Behavioral: Music Playing Task
- Order 2 (Experimental): Participants randomized to Order 2 will complete the four music playing tasks in the following order: (1) Improvisation, no live accompaniment (recorded accompaniment); (2) No improvisation (maintain beat), no live accompaniment (recorded accompaniment); (3) Improvisation, live accompaniment; (4) No improvisation (maintain beat), live accompaniment.
  Interventions: Behavioral: Music Playing Task
- Order 3 (Experimental): Participants randomized to Order 3 will complete the four music playing tasks in the following order: (1) No improvisation (maintain beat), live accompaniment; (2) Improvisation, live accompaniment; (3) No improvisation (maintain beat), no live accompaniment (recorded accompaniment); (4) Improvisation, no live accompaniment (recorded accompaniment).
  Interventions: Behavioral: Music Playing Task
- Order 4 (Experimental): Participants randomized to Order 3 will complete the four music playing tasks in the following order: (1) Improvisation, live accompaniment; (2) No improvisation (maintain beat), live accompaniment; (3) Improvisation, no live accompaniment (recorded accompaniment); (4) No improvisation (maintain beat), no live accompaniment (recorded accompaniment).
  Interventions: Behavioral: Music Playing Task

INTERVENTIONS:
Behavioral: Music Playing Task — For the music playing task, participants will tap on an MRI compatible MIDI drum in response to music, while following directions to either (1) maintain the beat of the music or (2) improvise a beat along with the music. Piano accompaniment for drum playing will be provided either (1) with a recording or (2) by a live music therapist. Participants will complete all four combinations of these music playing tasks following the sequence of experimental order 3. Each of the four tasks will be repeated with four one-minute songs, resulting in a total of 16 minutes of drum playing required to complete the study procedures. Participants will repeat the same task order with each song to facilitate task comprehension and task completion accuracy. Song order will be randomized for all participants.

SUMMARY:
This study will enroll stroke patients and healthy participants. Participants will complete baseline measures followed by a music playing task during fMRI and simultaneous measurement of motor response using electromyography (EMG) and accelerometry and affective response using electrodermal activity (EDA) and self-reports. The music task consists of tapping an MRI-compatible MIDI drum with either: (1) improvisation or maintaining the beat and (2) live or recorded piano accompaniment. The primary objectives are to identify the motor, affective, and neural outcomes of improvisation and live accompaniment in music playing tasks.

ELIGIBILITY:
Inclusion Criteria:

For participants with stroke, to be eligible to participate in this study, an individual must meet all the following criteria:

* hemiparesis resulting from a stroke (ischemic or hemorrhagic) at least 6 months before the enrollment into the study
* age from 18 to 89 years
* ability to move the wrist flexor and extensor muscles without help from the healthy side, scoring above 3 on the Medical Research Council (MRC) Scale for Muscle Strength, reflecting active movement against gravity
* no more than mild resistance to passive movement in the wrist extensor muscle - as demonstrated by a score <2 on the Ashworth Scale (Brashear et al.., 2002)
* a modified Rankin Scale (mRS) < 3 indicating moderate to mild disability and the ability to ambulate independently (Bonita & Beaglehole, 1988)
* ability to comprehend language and provide informed consent
* consenting to participate and willingness to complete MRI testing procedures

For neurologically normal control (NC) participants, to be eligible to participate in this study, an individual must meet all the following criteria:

* be matched for age, gender, and socioeconomic status (education level) to a previously enrolled participant with stroke
* age from 18 to 89 years
* no history of neurological injury
* ability to comprehend language and provide informed consent
* consenting to participate and willingness to complete MRI testing procedures

Exclusion Criteria:

* history of neurological injury other than stroke
* moderate to severe depression symptoms indicated by a score >10 on the Patient Health Questionnaire - 9 (PHQ-9; Koenke et al., 2001; Williams et al., 2005)
* visual impairment unable to be corrected with glasses/contact lenses sufficient to allow reading comprehension
* actively performing or practicing a musical instrument more than 2 hours/week
* musical anhedonia indicated by a score < 65 on the Barcelona Music Reward Questionnaire (BMRQ; Mas-Herrero et al., 2013)
* amusia as measured by the Montreal Battery of the Evaluation of Amusia (MBEA; Peretz et al., 2003)
* not being compatible with MRI testing, including having implanted devices, previous exposure to metallic fragments, large tattoos, claustrophobia, and pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Total Acceleration of Hand Movements during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using an MRI-compatible accelerometer attached to the hand with a Velcro strap.
Total Acceleration of Hand Movements during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using an MRI-compatible accelerometer attached to the hand with a Velcro strap.
Total Acceleration of Hand Movements during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using an MRI-compatible accelerometer attached to the hand with a Velcro strap.
Total Acceleration of Hand Movements during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using an MRI-compatible accelerometer attached to the hand with a Velcro strap.
Total Muscle Activation during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using MRI-compatible electromyography sensors placed on the arm.
Total Muscle Activation during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using MRI-compatible electromyography sensors placed on the arm.
Total Muscle Activation during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using MRI-compatible electromyography sensors placed on the arm.
Total Muscle Activation during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  This measurement will be taken using MRI-compatible electromyography sensors placed on the arm.
Neural Activation in Primary Motor Cortex during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.
Neural Activation in Primary Motor Cortex during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.
Neural Activation in Primary Motor Cortex during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.
Neural Activation in Primary Motor Cortex during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.
Neural Activation in Supplementary Motor Cortex during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.
Neural Activation in Supplementary Motor Cortex during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.
Neural Activation in Supplementary Motor Cortex during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.
Neural Activation in Supplementary Motor Cortex during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated.

SECONDARY OUTCOMES:
Electrodermal Activity (EDA) during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  EDA is a procedure for measuring emotional excitement by recording the skin's natural electrical activity. The measurements will be taken using two MRI-compatible sensors attached to the palm of the hand.
Electrodermal Activity (EDA) during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  EDA is a procedure for measuring emotional excitement by recording the skin's natural electrical activity. The measurements will be taken using two MRI-compatible sensors attached to the palm of the hand.
Electrodermal Activity (EDA) during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  EDA is a procedure for measuring emotional excitement by recording the skin's natural electrical activity. The measurements will be taken using two MRI-compatible sensors attached to the palm of the hand.
Electrodermal Activity (EDA) during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  EDA is a procedure for measuring emotional excitement by recording the skin's natural electrical activity. The measurements will be taken using two MRI-compatible sensors attached to the palm of the hand.
Music Playing Self-Report Questionnaire - Pleasure Score during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's pleasure while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater pleasure.
Music Playing Self-Report Questionnaire - Pleasure Score during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's pleasure while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater pleasure.
Music Playing Self-Report Questionnaire - Pleasure Score during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's pleasure while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater pleasure.
Music Playing Self-Report Questionnaire - Pleasure Score during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's pleasure while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater pleasure.
Music Playing Self-Report Questionnaire - Cognitive Challenge Score during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's cognitive challenge while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater cognitive challenge.
Music Playing Self-Report Questionnaire - Cognitive Challenge Score during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's cognitive challenge while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater cognitive challenge.
Music Playing Self-Report Questionnaire - Cognitive Challenge Score during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's cognitive challenge while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater cognitive challenge.
Music Playing Self-Report Questionnaire - Cognitive Challenge Score during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  The questionnaire includes 1 question measuring participant's cognitive challenge while performing the music activity. The item is rated on a Likert scale from 1 (low) to 5 (high); higher scores indicate greater cognitive challenge.
Neural Activation in Amygdala during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Amygdala during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Amygdala during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Amygdala during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventromedial Prefrontal Cortex during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventromedial Prefrontal Cortex during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventromedial Prefrontal Cortex during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventromedial Prefrontal Cortex during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventral Striatum during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventral Striatum during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventral Striatum during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Ventral Striatum during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Dorsolateral Prefrontal Cortex during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Dorsolateral Prefrontal Cortex during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Dorsolateral Prefrontal Cortex during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Neural Activation in Dorsolateral Prefrontal Cortex during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI).
Functional Connectivity with the Ventral Striatum during Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Psychophysiological interactions (PPI) analysis will be used with the seed in the ventral striatum.
Functional Connectivity with the Ventral Striatum during Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Psychophysiological interactions (PPI) analysis will be used with the seed in the ventral striatum.
Functional Connectivity with the Ventral Striatum during No Improvisation + No Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Psychophysiological interactions (PPI) analysis will be used with the seed in the ventral striatum.
Functional Connectivity with the Ventral Striatum during No Improvisation + Live Accompaniment Task | Day 1 (About 3 hours)
  Measured using functional MRI (fMRI). Psychophysiological interactions (PPI) analysis will be used with the seed in the ventral striatum.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Schambra, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: pripolles@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to pripolles@nyu.edu. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT06215703/ICF_000.pdf